CLINICAL TRIAL: NCT04034472
Title: Interdisciplinary Weight Loss Therapy Associate With the Use of Interactive Digital Technology as Adjuvant Tool to the Clinical Practices in Obesity
Brief Title: Interdisciplinary Weight Loss Therapy Associate With the Use of Interactive Digital Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana R. Damaso, Professor, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UNIFESP - GEO
Record Dates: First submitted 2019-03-15; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Obesity
Keywords: obesity; comorbidities; inflammation; digital technology; metabolic alterations
MeSH Terms: conditions — Obesity; Inflammation | interventions — Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiometabolic risk in women with obesity (Other): The use of interactive digital technology as adjuvant tool to the clinical practices in weight loss therapy emerges as an innovative strategy. However. it was note fully investigated if this can contribute to decrease inflammatory markers in obese women. In the present investigate it was amied to evaluate the effects of clinical approach associated to use of electronic means on inflammatory markers in women with obesity.
  Interventions: Other: Interdisciplinary intervention in obesity

INTERVENTIONS:
Other: Interdisciplinary intervention in obesity — Interdisciplinary weight loss intervention associate to the use of digital technology to treat obesity and related disorders

SUMMARY:
Obesity is a complex disease associate to metabolic alterations, which may lead to cardiometabolic risk in women with obesity. The use of interactive digital technology as adjuvante tool to the clinical practices in weight loss therapy emerges as an innovative strategy. However, it was note fully investigated if this kind of approach can contribute to improve inflammatory state and metabolic alterations in obese population.

DETAILED DESCRIPTION:
This study consists in a 12-week clinical interdisciplinary weight loss therapy, with endocrinologist, nutritionist, psychologist and exercise physiologist to evaluate the effects of clinical interdisciplinary therapy associated to use the eletronic means on inflammatory biomarkers and metabolic alterations in women with obesity.

The present study was composed by a sample of obese women (20 to 45 years old), recruited through advertisements in the media (newspapers, magazines, radio, television and social media - Twitter®, Facebook® and Instagram®). The volunteers lived in the city of São Paulo or nearby, so they could attend monthly the University on the days of the clinical, nutritional, psychological and exercise evaluations, counseling, educational sessions and motivational strategies supporting adherence. To complete the Education Behaviors Program the volunteers follow weekly the instructions found in the Platform #12Semanas®. All participants met the inclusion criteria for the obesity profile according to the World Health Organization (WHO), presenting Body Mass Index (BMI) values above 30 kg/m². Patients with any pathology that could compromise the results of the study (heart disease, musculoskeletal deformities, diseases related to the immune system, genetic, metabolic or endocrine diseases, identified by the physician) were not included in the study. Anthropometric measures, body composition by bio-impedance and bood samples were collected to serum analysis.

ELIGIBILITY:
Inclusion Criteria:

* obesity diagnosis;
* body mass index (BMI) values above 30 kg/m²
* adult
* aged 20-45 years

Exclusion Criteria:

* presence of heart diseases
* musculoskeletal deformities
* diseases related to the immune system

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
Body weight (kg) | 12 weeks
  Body weight was measured using light clothes and barefoot on a Filizola® scale to 0,1kg and capacity of 180kg.
Body Fat mass (kg) | 12 weeks
  Body fat mass was measured by Bio-impedance meter (BIA) by the device BIODYNAMICS 310e (TBW®).
Glucose Concentration | 12 weeks
  Blood samples were collected at the outpatient clinic at approximately 8:00 A.M. after an overnight fast (12h). Glucose concentration were available by commercial kits.
Body Lean mass (kg) | 12 weeks
  Body lean mass was measured by Bio-impedance meter (BIA) by the device BIODYNAMICS 310e (TBW®).
Basal Metabolic Rate (KJ/day) | 12 weeks
  Basal Metabolic Rate was estimated by Bio-impedance meter (BIA) - device BIODYNAMICS 310e (TBW®).
Insulin Concentration | 12 weeks
  Blood samples were collected at the outpatient clinic at approximately 8:00 A.M. after an overnight fast (12h). Insulin concentration were available by commercial kits. Insulin resistance was assessed using the homeostasis model assessment-insulin resistance (HOMA-IR). The cutoff value determined for Brazilian population is HOMA-IR>2.71 for classifying the subjects with insulin resistance.
Human Fibroblast Growth Factor 21 | 12 weeks
  Blood samples were collected at the outpatient clinic at approximately 8:00 A.M. after an overnight fast (12h). The assays of Human Fibroblast Growth Factor 21 (FGF-21) concentration were determined by ELISA.
Adiponectin | 12 weeks
  Blood samples were collected at the outpatient clinic at approximately 8:00 A.M. after an overnight fast (12h). The assays of adiponectin concentration were determined by ELISA.
Atrial Natriuretic Peptide | 12 weeks
  Blood samples were collected at the outpatient clinic at approximately 8:00 A.M. after an overnight fast (12h). The assays of atrial natriuretic peptide (ANP) concentration were determined by ELISA.
Leptin | 12 weeks
  Blood samples were collected at the outpatient clinic at approximately 8:00 A.M. after an overnight fast (12h). The assays of leptin concentration were determined by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No